CLINICAL TRIAL: NCT02610764
Title: Resectable Esophageal Adenocarcinoma: The Influence of Multimodal Therapy on the Prevalence and Enumeration of Circulating Tumor Cells in Comparison With Conventional Response Evaluation in a Feasibility Study
Brief Title: Pilot Sudy: Resectable Esophageal Adenocarcinoma and the Relevance of CTC
Acronym: ESO-CTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Dr. Birte Kulemann, Resident in Surgery, University Hospital Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ESO-CTC (Pilot)
Record Dates: First submitted 2015-11-15; First posted 2015-11-20 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Esophageal Adenocarcinoma
Keywords: Circulating Tumor Cells; Response evaluation
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Neoplastic Cells, Circulating | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental diagnostic test (Experimental): Evaluation and enumeration of circulating Tumor cells from the blood with two different CTC-detection platforms: one established test (CellSearch) and one experimental test (ScreenCell).
  Control diagnostic test: CT-Scan of the Chest and the Abdomen, Endoscopy and Endosonography, Clinical response and histo pathologic response. (% Of vital tumor Cells in the histologic specimen).
  Interventions: Procedure: Blood Test for CTC evaluation

INTERVENTIONS:
Procedure: Blood Test for CTC evaluation

SUMMARY:
To investigate the feasibility of evaluation of prevalence and clinical significance and relevance of circulating tumor cells (CTC) in the blood of patients with resectable adenocarcinoma of the esophagus (EAC) treated with multimodal therapy in a pilot study. The primary hypothesis is that the number of CTC correlates with tumor burden and response to treatment. One established and one experimental CTC detection platform will be investigated. Investigators will evaluate the prevalence and enumeration of CTC before neoadjuvant treatment (time point 1), after neoadjuvant treatment & before operation (time point 2) and after the operation (time point 3). Results will be compared with healthy controls (one time point) and correlated with conventional response to treatment evaluation. The persistent presence of CTC could be a marker for worse response to treatment and predict early recurrence.

DETAILED DESCRIPTION:
Little is known of the prevalence and clinical relevance of CTC in EAC, with the available data arising from heterogeneous patient populations using varied detection methods; but they are promising tools to improve staging and prediction of treatment response to perioperative and operative therapy.

The limited reports on resectable EAC use the epithelial-antibody dependent CellSearch method for CTC isolation and report a CTC-positivity rate of only 15-18% in non-pre-treated patients but with clinical relevance. It is thus needed to evaluate the relevance of CTC in the context of multimodal treatment courses.

This pilot study will investigate the CTC in the blood of patients with resectable EAC treated with multimodal therapy. Data on prevalence and enumeration of CTC will be generated. Two CTC isolation methods will be investigated, the established and expensive surface-antibody-dependent CellSearch method, and the antibody-independent and less expensive isolation by size (ISET; ScreenCell) method. The ISET method will additionally be investigated in healthy controls to get data on specificity.

The study can accomplish several goals through the use of two CTC detection platforms: 1) to determine the prevalence and number of CTC in resectable EAC under multimodal treatment, and 2) to investigate the potential role of CTC in predicting response to treatment and prognosis before neoadjuvant treatment, after neoadjuvant treatment and before operation as well as after the operation.

The primary hypothesis is that the enumeration of the CTC correlates with tumor burden and will reflect the response to treatment. To date the response to treatment is assessed with a combination of CT-morphologic, endoscopic, clinical (dysphagia) and finally histology. This assessment is used as control.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma of the esophagus According to the UICC definition (TNM7),
* pre-treatment stage cT1N+, M0 or cT2-4aN0/N+, M0 ,
* Age≥18 years,
* scheduled for a multimodal therapeutic concept.

Exclusion Criteria:

* Tumors of squamous, adenosquamous or other non-adenocarcinoma histology, patients with advanced inoperable or metastatic esophageal adenocarcinoma.
* Esophageal adenocarcinoma cT1N0 and cT4b,
* Gastric carcinoma.
* Prior chemotherapy for gastrointestinal cancer. Clinically not eligible for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change of numbers of CTCs in patients with resectable EAC at diagnosis, after neoadjuvant treatment and after surgery. | 1 year

SECONDARY OUTCOMES:
Number of patients with detectable CTCs at diagnosis, after neoadjuvant treatment and after surgery. | 1 year
  Number of patients with detectable CTCs isolated with the ISET device compared to the CellSearch method.

OTHER OUTCOMES:
Overall survival | 2 years after recruitment of last patient
  The overall survival will be correlated with the number of CTC at the different timepoints.
Progression free survival | 2 years after recruitment of last patient
  The progression free survival will be correlated with the number of CTC at the different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Birte Kulemann, Dr. med., Principal Investigator — University Hospital Freiburg
Locations (1):
- University of Freiburg - Medical Center, Freiburg im Breisgau, Baden-Würtemberg, Germany